CLINICAL TRIAL: NCT03876509
Title: Non-invasive Diagnosis of Pulmonary Hypertension by Thoracic Impedance Cardiography - a Prospective Study
Brief Title: Non-invasive Diagnosis of Pulmonary Hypertension by Impedance Cardiography
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 29-478 ex 16/17
Record Dates: First submitted 2018-12-05; First posted 2019-03-15 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Hypertension
Keywords: impedance cardiography
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Cardiography, Impedance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Impedance Cardiography: Impedance Cardiography
  Interventions: Diagnostic Test: Impedance Cardiography

INTERVENTIONS:
Diagnostic Test: Impedance Cardiography — Impedance Cardiography will be conducted in patients with suspected Pulmonary Hypertension within an interval of 24 hours to right-heart catheterization. Usually, 8 electrodes will be attached on the neck and thorax of the patient. These electrodes will produce current (max 400µA) and measure the voltage which is produced by the current running through the body. The Signal will be analyzed for specific signs of Pulmonary Hypertension.
  At the same time electrocardiography and non-invasive continuous blood pressure will be measured.

SUMMARY:
The goal of the study is to prospectively evaluate Impedance Cardiography as a tool to detect pulmonary hypertension. According to our hypothesis Impedance Cardiography is a valuable method to differentiate patients without pulmonary hypertension from patients with pulmonary hypertension. The main objective is to determine the sensitivity and specificity in comparison to the gold standard right heart catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Patients with clinical indication for right heart catheterization

Exclusion Criteria:

* known Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the clinical department of Pulmonology of the Medical University of Graz undergoing right heart catheterization for clinical reasons will be included
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Diagnosis of pulmonary hypertension | 1 hour
  The sensitivity and specificity of Impedance Cardiography in the diagnosis of pulmonary Hypertension (as compared with the Gold Standard right heart catheterization) will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Division of Pulmonology, Graz, Styria, Austria